CLINICAL TRIAL: NCT06598033
Title: Vitamin C Plus Cordyceps to Quality of Life in Patients With Terminal Stage Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-13
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Phytotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VC plus herbal medicine (Experimental): Vitamin C 300 mg/day, TID, PO. Reishi, 2 g/day, BID, PO. Cordyceps, 2 g/day, BID, PO.
  Interventions: Drug: VC plus herbal medicine

INTERVENTIONS:
Drug: VC plus herbal medicine — Vitamin C 300 mg/day, TID, PO. Reishi, 2 g/day, BID, PO. Cordyceps, 2 g/day, BID, PO.

SUMMARY:
The purpose of this study is to evaluate the efficacy of vitamin C plus herbal medicine in improving the quality of life for metastatic pancreatic cancer patients who are resistant to chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. In 2011, the PRODIGE trial has shown that oxaliplatin, irinotecan, fluorouracil, and leucovorin (FOLFIRINOX) was associated with a survival advantage but had increased toxicity. In 2013, the MPACT trial has confirmed the efficacy of gemcitabine combined with nab-paclitaxel as the first-line treatment to metastatic pancreatic cancer. However, the side-effects related to chemotherapy including anemia, hand/foot numbness, fatigue, nausea, and malnutrition have impaired the quality of life for patients.

Vitamin C, also called ascorbate, is an essential nutrient for the human body. It modulates metabolism, immune reaction, collagen synthesis, and iron absorption. Some studies have shown that high-dose intravenous Vitamin C may be effective against various types of cancer. Meanwhile, medium or low dose of Vitamin C may increase iron absorption, improve anemia, alleviate pain and hand/foot numbness, and thus improve the quality of life for patients with terminal stage pancreatic cancer. In addition, numerous evidence has proved the efficacy of Reishi and Cordyceps in alleviating the side effects related to chemotherapy.

The purpose of this study is to evaluate the efficacy of vitamin C plus herbal medicine on improving the quality of life for metastatic pancreatic cancer patients who are resistant to two lines of systemic chemotherapy, including gemcitabine based, fluorouracil based, or other regimen. Fifty patients who have tumor progression after receiving two lines of chemotherapy will be recruited. These patients will receive Vitamin C plus herbal medicine. Quality of life, rate of hand/foot numbness, severity of pain, rate of anemia, and overall survival are measured.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to understand and the willingness to sign a written informed consent document.

  * Age ≥ 18 years and ≤ 80 years.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
  * Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
  * Tumor progression after two lines of treatments.
  * Adequate organ performance based on laboratory blood tests.
  * Presence of at least of one measurable lesion in agreement to RECIST criteria.
  * The expected survival ≥ 1 months.
  * Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* • The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.

  * Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
  * Pregnant or nursing women.
  * Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
  * Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
  * Renal insufficiency or dialysis
  * Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
  * Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) questionnaire | 1 month
  Change of QOL after every cycle of treatment using ORTC QLQ-C30 (version 3). Scale 1-7, higher scores mean a better outcome.

SECONDARY OUTCOMES:
Rate of hand-foot skin reaction, HFSR | 1 month
  Rate of HFSR after every cycle of treatment
Rate of anemia | 1 month
  Rate of anemia after every cycle of treatment
Overall survival，OS | 1 month
  OS of subjects from recruiting to the time of death from any cause
Change of numeric rating scale (NRS) | 1 month
  Change of numeric rating scale (NRS) and the administration of analgesic drugs after every cycle of treatment. NRS scale 0-10. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Principal Investigator — Shanghai Cancer Center
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Das G, Shin HS, Leyva-Gomez G, Prado-Audelo MLD, Cortes H, Singh YD, Panda MK, Mishra AP, Nigam M, Saklani S, Chaturi PK, Martorell M, Cruz-Martins N, Sharma V, Garg N, Sharma R, Patra JK. Cordyceps spp.: A Review on Its Immune-Stimulatory and Other Biological Potentials. Front Pharmacol. 2021 Feb 8;11:602364. doi: 10.3389/fphar.2020.602364. eCollection 2020. PMID 33628175
- [Background] Wang X, Zhu X, Liu Y, Liu H, Xiao Z, Luo G. Efficacy of vitamin C on chemotherapy-related anemia in pancreatic cancer: study protocol for a randomized controlled trial. Trials. 2024 Jul 29;25(1):512. doi: 10.1186/s13063-024-08345-w. PMID 39075587
- [Background] Sohretoglu D, Huang S. Ganoderma lucidum Polysaccharides as An Anti-cancer Agent. Anticancer Agents Med Chem. 2018;18(5):667-674. doi: 10.2174/1871520617666171113121246. PMID 29141563